CLINICAL TRIAL: NCT04324099
Title: Investigating the Specificity of Neural Correlates for Emotion Processing Deficits in Conduct Disorder and Autism Spectrum Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-02386;pk17Stadler
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Autism-Spectrum Disorder; Conduct Disorder
Keywords: Callous-Unemotional traits; emotion processing deficits; dysfunctional cognitive control processes
MeSH Terms: conditions — Child Development Disorders, Pervasive; Conduct Disorder | interventions — Surveys and Questionnaires; Childhood Trauma Questionnaire; Vorinostat; BES; Intensive Care Units; Spermine Synthase

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conduct disorder: children and adolescents with CD
  Interventions: Other: neuroimaging session (with simultaneously acquired eye-tracking); Other: Questionnaire (for children) assessing traumatic experiences (Childhood trauma questionnaire (CTQ)); Other: Social and Health Assessment (SAHA) questionnaire (for children); Other: Massachusetts Youth Screening Instrument (MAYSI-2) (for children); Other: Interpersonal Reactivity Index (IRI) (for children); Other: Youth Psychopathic Traits Inventory (YPI) (for children); Other: Reactive Proactive Questionnaire (RPQ) (for children); Other: Emotion Regulation Questionnaire (for children); Other: Basic Empathy Scale (BES) (for children); Other: Pubertal Development Scale (PDS) (for children); Other: Alabama Parenting Questionnaire (APQ) (for parents); Other: Inventory of Callous Unemotional Traits (ICU) (for parents); Other: Child Behavior Checklist (CBCL) (for parents); Other: Griffith Empathy Measure (GEM) (for parents); Other: Social Responsiveness Scale (SRS) (for parents)
- Autism-Spectrum disorder: children and adolescents with ASD
  Interventions: Other: neuroimaging session (with simultaneously acquired eye-tracking); Other: Questionnaire (for children) assessing traumatic experiences (Childhood trauma questionnaire (CTQ)); Other: Social and Health Assessment (SAHA) questionnaire (for children); Other: Massachusetts Youth Screening Instrument (MAYSI-2) (for children); Other: Interpersonal Reactivity Index (IRI) (for children); Other: Youth Psychopathic Traits Inventory (YPI) (for children); Other: Reactive Proactive Questionnaire (RPQ) (for children); Other: Emotion Regulation Questionnaire (for children); Other: Basic Empathy Scale (BES) (for children); Other: Pubertal Development Scale (PDS) (for children); Other: Alabama Parenting Questionnaire (APQ) (for parents); Other: Inventory of Callous Unemotional Traits (ICU) (for parents); Other: Child Behavior Checklist (CBCL) (for parents); Other: Griffith Empathy Measure (GEM) (for parents); Other: Social Responsiveness Scale (SRS) (for parents)
- typically developing adolescents: typically developing adolescents
  Interventions: Other: neuroimaging session (with simultaneously acquired eye-tracking); Other: Questionnaire (for children) assessing traumatic experiences (Childhood trauma questionnaire (CTQ)); Other: Social and Health Assessment (SAHA) questionnaire (for children); Other: Massachusetts Youth Screening Instrument (MAYSI-2) (for children); Other: Interpersonal Reactivity Index (IRI) (for children); Other: Youth Psychopathic Traits Inventory (YPI) (for children); Other: Reactive Proactive Questionnaire (RPQ) (for children); Other: Emotion Regulation Questionnaire (for children); Other: Basic Empathy Scale (BES) (for children); Other: Pubertal Development Scale (PDS) (for children); Other: Alabama Parenting Questionnaire (APQ) (for parents); Other: Inventory of Callous Unemotional Traits (ICU) (for parents); Other: Child Behavior Checklist (CBCL) (for parents); Other: Griffith Empathy Measure (GEM) (for parents); Other: Social Responsiveness Scale (SRS) (for parents)

INTERVENTIONS:
Other: neuroimaging session (with simultaneously acquired eye-tracking) — neuroimaging session, including two functional neuroimaging paradigms (ca. 15-20 minutes each) and a short structural image acquisition (mprage) for coregistration. Functional Magnetic Brain Imaging (fMRI) and simultaneous eye-tracking data will be collected during the paradigms: 1) an emotion processing paradigm (adapted from Passamonti et al., 2010); and 2) an emotional Go/noGo paradigm (adapted from Hare et al., 2008).
Other: Questionnaire (for children) assessing traumatic experiences (Childhood trauma questionnaire (CTQ)) — The Childhood Trauma Questionnaire is a brief survey of six early traumatic experiences (death, divorce, violence, sexual abuse, illness or other), and assesses individual's understanding of their childhood trauma.
Other: Social and Health Assessment (SAHA) questionnaire (for children) — Self reported survey assessing social and mental health with four aspects of parenting determined (parental involvement, parental warmth, parental control, and inconsistency of parenting).
Other: Massachusetts Youth Screening Instrument (MAYSI-2) (for children) — The Massachusetts Youth Screening Instrument (MAYSI-2) is a screening instrument developed for detecting mental health needs in youth aged 12-17. Designed as a low-cost, easily administered tool, it screens for multiple issues and can be administered in 10-15 minutes. It is divided into seven scales composed of 52 questions that are designed to detect alcohol/drug use, angryirritable behavior, depression-anxiety, somatic complaints, suicide ideation, thought disturbance, and traumatic experience. Youths answer YES or NO concerning whether each item has been true for them "within the past few months.
Other: Interpersonal Reactivity Index (IRI) (for children) — The Interpersonal Reactivity Index is a measure of dispositional empathy that takes as its starting point the notion that empathy consists of a set of separate but related constructs. The instrument contains four seven-item subscales (seven Likert items each), each tapping a separate facet of empathy (Empathic Concern, Perspective Taking, Personal Distress, and Fantasy). The 28-item IRI contains four subscales
Other: Youth Psychopathic Traits Inventory (YPI) (for children) — self-report screening measures to assess psychopathic traits in youth assessing 10 core personality traits associated with the construct (grandiosity, lying, manipulation, callousness, unemotionality, impulsivity, irresponsibility, dishonest charm, remorselessness, and thrill seeking). Each item is scored on an ordinal 4-point Likert scale (1 = Does not apply at all, to 4 = Applies very well). Higher scores reflect an increased presence of psychopathic traits.
Other: Reactive Proactive Questionnaire (RPQ) (for children) — The Reactive-Proactive Questionnaire (RPQ) scores (0 (never), 1 sometimes, 2 (often)) for proactive aggression items and reactive items. Proactive and reactive scale scores are summated to obtain total aggression scores.
Other: Emotion Regulation Questionnaire (for children) — 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree)
Other: Basic Empathy Scale (BES) (for children) — The Basic Empathy Scale (BES) measures 20 items (affective and cognitive empathy) on a Five-point Likert-type scale.
Other: Pubertal Development Scale (PDS) (for children) — self-report measure of physical development which has been shown to be correlated with measures of pubertal development derived from physical examination. Responses are coded on 4-point scales (1 = no development and 4 = completed development). For girls, a yes-no question about onset of menarche is weighted more heavily (1 = no and 4 = yes). For both genders, ratings are then averaged to create an overall score for physical maturation.
Other: Alabama Parenting Questionnaire (APQ) (for parents) — The APQ measures five dimensions of parenting that are relevant to the etiology and treatment of child externalizing problems: (1) positive involvement with children, (2) supervision and monitoring, (3) use of positive discipline techniques, (4) consistency in the use of such discipline and (5) use of corporal punishment (42 self-reported responses, rated on a 5-point Likert scale- 1 (never) to 5 (always) for both child and parent forms)
Other: Inventory of Callous Unemotional Traits (ICU) (for parents) — 24-item questionnaire designed to provide a comprehensive assessment of callous and unemotional traits.The ICU has three subscales: Callousness, Uncaring, and Unemotional. The ICU is made up of statements with a 4-point Likert scale, ranging from 0 (Not at all true) to 3 (Definitely True), with higher scores indicating greater CU traits.
Other: Child Behavior Checklist (CBCL) (for parents) — The eight empirically-based syndrome scales are:
  1. Aggressive Behavior
  2. Anxious/Depressed
  3. Attention Problems
  4. Rule-Breaking Behavior
  5. Somatic Complaints
  6. Social Problems
  7. Thought Problems
  8. Withdrawn/Depressed. Higher scores indicate greater Problems.
Other: Griffith Empathy Measure (GEM) (for parents) — self-report 23-item measure of empathy in which the respondent answers each item on a nine-point Likert scale from strongly disagree to strongly agree
Other: Social Responsiveness Scale (SRS) (for parents) — Social Responsiveness Scale (SRS) measures social ability of children from 4 years to 18 years old. It is used primarily with individuals with Autism Spectrum Disorder (ASD), family members of individuals with ASD, and others who have social impairments. Parent or teacher questionnaire (65 items on a 4-point Likert scale). High scores are associated with more severe social impairments.

SUMMARY:
This study is

1. to investigate the differential and shared neural underpinnings of facial emotion processing within Conduct disorder (CD) and Autism-Spectrum disorder (ASD) and
2. to investigate the interaction between deficits in emotion processing and dysfunctional cognitive control processes.

Differences in emotion processing and the underlying neural underpinnings of such differences will be assessed by means of functional magnetic resonance imaging (fMRI) without any contrast agent, combined with adapted emotion processing paradigms and eye tracking techniques.

ELIGIBILITY:
Inclusion Criteria:

* For all participants: age between 10 and 18 years and an intelligence quotient score of 70 or higher.
* For patient groups: confirmed clinical diagnoses according to Diagnostic and Statistical Manual (DSM)-5 of CD or ASD (depending on the group), without comorbid depression or anxiety psychological disorders.

Exclusion Criteria:

* For all participants: low intelligence (IQ<70, as they might otherwise not fully understand what they are expected to do inside the scanner), insufficient German language skills or any contraindications for MRI (e.g. pregnancy, any non-removable metal within the subjects' body, claustrophobia).
* For patient groups: severe developmental disorders, comorbid depressive and/or anxiety disorders will also be excluded from the study since it was shown that these patients might have problems in attention allocation under emotional stimulation.
* For typically developing participants: suspicion of an undiagnosed clinical disorder

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: German speaking children and adolescents (10-18 years of age) attended at the Kinder- und Jugendpsychiatrischen Klinik Basel (KJPK) and with a confirmed diagnosis of CD or ASD.
  Typically developing children will be recruited using leaflets (will be distributed in the KJPK clinics and in socioeconomically diversesecondary schools within the Canton of Basel-Stadt).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
difference between groups (children and adolescents with CD, ASD and typically developing adolescents) in neural activity | fMRI imaging Day 1
  difference between groups in neural activity as measured by Blood Oxygen Level Dependent (BOLD) signal during emotion processing using a priori defined regions of interest (ROIs) including the insula, amygdala, and ventromedial prefrontal Cortex in fMRI

SECONDARY OUTCOMES:
Emotion processing task (fMRI) | fMRI imaging Day 1
  Emotion processing task (fMRI): measures of eye gaze collected by eye-tracking

CONTACTS AND LOCATIONS:
Overall Officials: Christina Stadler, Prof. Dr. med, Principal Investigator — Department of Child and Adolescent Psychiatry, KJPK (UPK)
Locations (1):
- Department of Child and Adolescent Psychiatry, KJPK (UPK), Basel, Switzerland